CLINICAL TRIAL: NCT04364568
Title: Minor Traumatic Brain Injury : MRI Examination of Consequences and Social Insertion
Acronym: TRACE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty recruiting and no sociologists
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Regional Council of Auvergne-Rhône-Alpes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 38RC19.305
Record Dates: First submitted 2020-03-20; First posted 2020-04-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Magnetic Resonance Spectroscopy; Interview, Psychological

STUDY DESIGN:
Intervention Model Description: prospective, monocentric, etiological cohort study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic group at three month (Experimental): Rivermead Post-Concussion Syndrome >= 12 MRI and clinical exam and sociological interview at day 105 (+/-15 days) 6 months follow up : sociological interview
  1 year follow up : psychological and sociological interview, Rivermead Post Concussion Syndrome questionnaire
  Interventions: Radiation: Magnetic Resonance Imaging
- Asymptomatic group at three month (Experimental): Rivermead Post-Concussion Syndrome < 12 MRI and clinical exam and sociological interview at day 105 (+/-15 days) 6 months follow up : sociological interview
  1 year follow up : psychological and sociological interview, Rivermead Post Concussion Syndrome questionnaire
  Interventions: Radiation: Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging — IRM Sequences T1, T2, FLAIR, T2*, Cerebral Blood Flow (CBF) et mean diffusivity (MD)
  Other Names: Sociological interview; Psychological interview

SUMMARY:
Minor traumatic brain injury (mTBI) (Glasgow Coma Scale 13 to 15) represent 70 to 90% of traumatic brain injury. Different disorders may occur after a traumatic minor brain injury (somatic, cognitive or affective) within 2 weeks.

For 10 to 20% these symptoms are persistent and are part of post-concussion syndrome. Today a small amount of tools to predict this syndrome are available. Cerebral CT scan, a routine test for mTBI, isn't relevant to predict the post concussion syndrome.

In order to improve understanding of the evolution toward this complication, it seems relevant to run a multimodal study.

Multiparameter MRI combined to psychological and sociological evaluations cold provide a better global perception.

ELIGIBILITY:
Inclusion Criteria:

* Patients who answered to psychological questionnaires 3 month after mTBI
* Patients with mTBI according to European Federation of Neurological Societies
* Initial CT scan indication according to 2012 French Society of Emergency Medicine and European Federation of Neurological Societies
* Health insurance
* Written consent

Exclusion Criteria:

* Under 18 years
* Psychiatric or neurologic history with long term treatment
* Hospitalization due to extra-cranial wounds or intoxication (except alcool)
* MTBI due to aggression
* MRI contraindication
* Inability to understand french language
* Pregnant or breastfeeding women
* Incapacitated patients in accordance with article L 1121-5 to L1121-8 of the public health code
* Patients in another study's exclusion time
* Inability to have a follow-up
* Patients who can't be reached in case of emergency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Compare the mean lesion volume fraction found in multiparametric magnetic resonance imaging between patients with and without post-concussions syndrome, three months after a mild Traumatic Brain Injury. | 3 months
  Mean of cerebral volume fraction corresponding to lesions areas, found in multiparametrical magnetic resonance imaging (expressed as a percentage), 3 months after mild traumatic brain injury.

SECONDARY OUTCOMES:
Describe correlation between anamnestic risk factors, demographic data and post-concussion syndrome occurence | 3 months
  Describe correlation between risk factor and the development of post-concussion syndrome.
  Describe risk factors as demographic factors and medical history correlated with the development of post-concussion syndrome.
  The risk factors studies will be:
  * Age (median in years)
  * Sex
  * Cohabitation status
  * Education
  * Daily consumption of alcohol
  * Smoking
  * Glasgow score
  * Loss of consciousness after the trauma
  * Associated injuries This information will be obtained using the medical record and by interviewing the patient. The presence of post-concussion syndrome will be defined using the Rivermead Post-concussion Symptoms Questionnaire. The presence of post-concussion syndrome will correspond to a score higher than 12.
Level of asymmetry of the signal between each hemisphere, for each magnetic resonance imagings equence, and with the techniques of ROI (Regions of Interests): asymmetry threshold corresponding to a lesion. | 3 months
  Measuring the level of asymmetry of the signal between each hemisphere, for each magnetic resonance imaging sequence, and with the techniques of ROI (Regions of Interests) ;to determine the asymmetry threshold corresponding to a lesion.
Graph metrics in resting-state functional magnetic resonance imaging in both groups | 3 months
  Describe the graph metrics in resting-state functional MRI in both groups
Clinical correlation of magnetic resonance imaging with symptoms. | 3 months
  Look for a clinical correlation between psychological evaluation tests and magnetic resonance imaging observations such as damages zones.
Describe in both groups, the evolution of symptomatology at one year | 12 months
  Describe in both groups, the evolution of symptomatology at one year with the Rivermead Post-Concussion Syndrome Questionnaire (RPCSQ). The Rivermead questionnaire ranges from 0 to 64. The presence of post-concussion syndrome will correspond to a score higher than 12.
Evaluate the impact of mTBI on patients' lifestyles | 6 months
  Sociologic interview to understand the impact of mTBI on patients' lifestyles and social insertion.
Evaluate the impact of mTBI on patients' lifestyles | 12 months
  Sociologic interview to understand the impact of mTBI on patients' lifestyles and social insertion.
Evaluate the impact of social characteristics at stake and the resources mobilized | 6 months
  Understand the impact of social characteristics at stake and the resources mobilized in the social life's re-establishment post TBI through a sociologic interview
Evaluate the impact of social characteristics and the resources mobilized | 12 months
  Understand the impact of social characteristics at stake and the resources mobilized in the social life's re-establishment post TBI through a sociologic interview
Evaluate the experience of mTBI and post-concussion syndrome through the patient's personal appreciation, the judgement of family and friends and the medical follow-up of the general practitioner. | 6 months
  Sociologic questionnaires to different actors of the patient recovery to understand the experience of mTBI and post-concussion syndrome :
  * the patient's personal appreciation,
  * the judgement of family and friends
  * the medical follow-up of the general practitioner.
Evaluate the experience of mTBI and post-concussion syndrome through the patient's personal appreciation, the judgement of family and friends and the medical follow-up of the general practitioner. | 12 months
  Sociologic questionnaires to different actors of the patient recovery to understand the experience of mTBI and post-concussion syndrome :
  * the patient's personal appreciation,
  * the judgement of family and friends
  * the medical follow-up of the general practitioner.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided